CLINICAL TRIAL: NCT04345159
Title: Association Between Long-term Hydroxychloroquine Treatment and Outcome of a History of Symptoms Suggestive of COVID-19 Infection During the Epidemic Period in France in Patients With Autoimmune Disease
Acronym: COVCALL
Status: Completed | Type: Observational
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: GDE_2020_11
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2021-01-07 (Actual); Status verified 2021-01

CONDITIONS: SARS-CoV-2; Systemic Lupus Erythematosus; Rheumatoid Arthritis; Sjogren's Syndrome; Psoriatic Arthritis
Keywords: Hydroxychloroquine
MeSH Terms: conditions — Lupus Erythematosus, Systemic; Arthritis, Rheumatoid; Sjogren's Syndrome; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with autoimmune disease: Selected using appropriate keywords in the Foundation Rothschild Hospital EMR, consenting to participate in the study.
  Interventions: Other: Questionnaire by phone call

INTERVENTIONS:
Other: Questionnaire by phone call — 2 questionnaires : at inclusion and 4 months later. The exposure to hydroxychloroquine and the history of autoimmune disease is determined during the phone call along with other exposure factors. The symptoms presented by the patient are classified in "Suggestive of a COVID-19 infection" or "Not suggestive of COVID-19 infection" by a team of internists and infectious diseases specialists, by studying the questionnaires after the completion in a blind-manner regarding the hydroxychloroquine intake.

SUMMARY:
This epidemiological, transversal, cohort study aims to determine the potential influence of an active long-term hydroxychloroquine intake over the prevalence of a history of symptoms evocative of a COVID-19 infection in patients with a history of systemic lupus erythematosus, rheumatoid arthritis, Sjogren's syndrome or psoriatic arthritis, during the epidemic period in France. The information is gathered using a standardized questionnaire, by phone call.

ELIGIBILITY:
Inclusion Criteria:

* History of Systemic Lupus Erythematosus, Rheumatoid arthritis, Sjogren's Syndrome or Psoriatic Arthritis.

Exclusion Criteria:

* beginning, or end, of an hydroxychloroquine treatment between Jan 1, 2020 and day of the phone call.
* Bad treatment compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen at least one time at Rothschild Foundation with history of Systemic Lupus Erythematosus, Rheumatoid arthritis, Sjogren's Syndrome, Psoriatic Arthritis.
Sampling Method: Non-Probability Sample
Enrollment: 572 (Actual)
Dates: Start 2020-04-17 (Actual); Primary Completion 2020-11-30 (Actual); Study Completion 2020-11-30 (Actual)

PRIMARY OUTCOMES:
Adjusted Odds Ratio | 4 months after inclusion
  Adjusted Odds Ratio measuring the association between an exposure to long-term hydroxychloroquine intake and a history of symptoms compatible with a COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume DEBELLEMANIERE, MD, Principal Investigator — Fondation Adolphe de Rothschild
Locations (1):
- Fondation Adolphe de Rothschild, Paris, France

REFERENCES:
- [Derived] Guillaume D, Magalie B, Sina E, Imene SM, Frederic V, Mathieu D, Aurore M, Yoni G, Emma E, Charlotte B, Laura F, Alain S, Steven N, Pierre Z, Jean-Luc F, Romain C, Alice GD, Adrien M, Wassim G, Pierre-Emmanuel R, Christophe P, Catherine C, Kevin B, Thomas S, Damien G. Antirheumatic Drug Intake Influence on Occurrence of COVID-19 Infection in Ambulatory Patients with Immune-Mediated Inflammatory Diseases: A Cohort Study. Rheumatol Ther. 2021 Dec;8(4):1887-1895. doi: 10.1007/s40744-021-00373-1. Epub 2021 Sep 16. PMID 34529226